CLINICAL TRIAL: NCT04352010
Title: Therapy Online Plus (TOP+) - Comparing Two Online Interventions ("REMOTION" Resp. "Res-Up!") for Dealing With Challenging Life Circumstances
Brief Title: Therapy Online Plus (TOP+) - Comparing Two Online Interventions for Dealing With Challenging Life Circumstances
Acronym: TOP+
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ulrike Willutzki (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, Ulrike Willutzki, Professor, Clinical Psychology and Psychotherapy, University of Witten/Herdecke
Organization: University of Witten/Herdecke (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221/2019
Record Dates: First submitted 2020-03-25; First posted 2020-04-17 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Mental Disorders; Online-Intervention
Keywords: Internet-based Therapy; Resilience; Emotion Regulation; Outcome Research; Strengths; Psychotherapy
MeSH Terms: conditions — Mental Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online-Intervention "Res-Up!" (Experimental): Participants in the Res-Up! group get access to Res-Up! while waiting for psychotherapy or in addition to psychotherapy. Participants will answer questionnaires after inclusion as well as six and twelve weeks later.
  Interventions: Behavioral: Res-Up!
- Online-Intervention "REMOTION" (Experimental): Participants in the REMOTION group get access to REMOTION while waiting for psychotherapy or in addition to psychotherapy. Participants will answer questionnaires after inclusion as well as six and twelve weeks later.
  Interventions: Behavioral: REMOTION
- Wait-control group (Experimental): Participants in the wait-control group will not get access to the online-tools while waiting for psychotherapy or while in psychotherapy. Participants will answer questionnaires after inclusion, six weeks later and twelve weeks later.They get access to one of the online-tools after 12 weeks.
  Interventions: Other: Wait-Control Group

INTERVENTIONS:
Behavioral: Res-Up! — Res-Up! is an internet-based intervention focusing on patients' strengths and positive experiences that have effects on distress, protective factors and quality of life. The intervention is based on the Personal Model of Resilience (PMR; Padesky and Mooney, 2012), which is a positive intervention that utilizes patients' strengths to overcome problems.The PMR activates resilient emotions, thoughts, metaphors, images and behaviors in four steps during five sessions about the aquisition of resilient strategies and their use in daily life. A variety of elements based on different psychotherapy approaches (Cognitive Behavioral Therapy, Emotion Focused Therapy, Positive Therapy etc.) are integrated in the program. Participants should work through one module per week. The intervention is conducted as I-CBT via the platform Minddistrict.Res-Up! is administered as a standalone or an add-on treatment to psychotherapy.
  Arms: Online-Intervention "Res-Up!"
Behavioral: REMOTION — REMOTION is an internet-based intervention aimed at transdiagnostically reducing symptom severity and improving emotion regulation of psychotherapy patients. The structure of REMOTION is based on the idea of an extended process model of emotion regulation as postulated by J.J. Gross (2015). The program includes the following modules: introduction, psychoeducation, identification, selection, implementation and modification. A variety of elements based on different psychotherapy approaches (Cognitive Behavioral Therapy, Emotion Focused Therapy, Dialectical Behavior Therapy etc.) are integrated in the program. Participants should work through one module per week. REMOTION is administered as a standalone or an add-on treatment to psychotherapy.
  Arms: Online-Intervention "REMOTION"
Other: Wait-Control Group — In the waiting control group participants will answer questionnaires and they will gain access to either REMOTION or Res-Up! after twelve weeks.
  Arms: Wait-control group

SUMMARY:
Psychotherapy interventions can roughly be grouped into compensation-oriented strategies (compensating for and and modifying personal deficits of patients) versus capitalization-oriented strategies (building on patients' personal strengths). Improvement of emotion regulation (compensation-oriented) as well as the activation of resilience (capitalisation-oriented) have been identified as important transdiagnostic factors in the treatment of mental disorders. The study aims to compare compensation vs. capitalization strategies by using two online programs, centered either on emotion-regulation ("REMOTION") or on activating resilience ("Res-Up!"). Res-Up! and REMOTION are administered as stand-alone intervention or as add-on treatment to standard psychotherapy.

Participants will be randomly assigned to three study conditions (Res-Up!, REMOTION, waiting control group). Outcomes are assessed at baseline, after six weeks and after twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a mental disorder according to DSM-5
* Recruited at the training centers of the German Association for Behavior Therapy (Deutsche Gesellschaft für Verhaltenstherapie, DGVT) at Muenster, Bielefeld and Dortmund or at the Center of Mental Health and Psychotherapy, Witten/Herdecke University (all outpatients clinics

Exclusion Criteria:

* Insufficient German language skills
* Current severe episode of major depression
* Psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change on Brief Symptom Inventory - short form (BSI-18) over multiple time points | Change from Baseline, then after six weeks and after twelve weeks
  Franke, 2000; Internationally used self-report of symptom severity of patients [18 items] that includes three symptom scales, each including six items: Somatization, Depression, and Anxiety. Each measured on a 5-point scale according to how much one has been bothered by the symptom in the prior week.

SECONDARY OUTCOMES:
Change on Patient Health Questionnaire-9 (PHQ-9) over multiple time points | Baseline, then after six weeks and after twelve weeks
  Kroenke, Spitzer, & Williams, 2001; Internationally used self-report for screening, diagnosing, monitoring and measuring the severity of depression [9 items, 4-point scale ("not at all" to "nearly every day")]. It is the major depressive disorder module of the full PHQ.
Change on Witten Resource Questionnaire (WIRF) over multiple time points | Change from Baseline, then after six weeks and after twelve weeks
  Schürmann et al., 2019; Self-report of personal and external resources [37 items, 6-point Likert scale ("strongly disagree" to "strongly agree")]. Resources are measured in the three contexts: "everyday life", "crises well coped with" and "current problems" each including three subscales (action regulation, relaxation and social support).
Change on Rosenberg-Self-Esteem Scale (RSES) over multiple time points | Change from Baseline, then after six weeks and after twelve weeks
  Ferring & Filipp, 1996; Self-report of general self-esteem [10 items, 4-point scale ("strongly disagree" to "strongly agree")]. A total score will be computed with summed item scores (range: 0-30).
Change on Connor-Davidson Resilience Scale (CD-RISC-10) over multiple time points | Change from Baseline, then after six weeks and after twelve weeks
  Sarubin et al., 2015; Internationally used self-report of individual resilience [short version: 10 items, each rated on a 5-point scale (0-4), with higher scores reflecting stronger resilience]. A total score will be computed with averaged item scores.
Change on Self-assessment of Emotion Regulation Skills (Selbsteinschätzung emotionaler Kompetenzen; SEK-27) over multiple time points | Change from Baseline, then after six weeks and after twelve weeks
  Berking & Znoj, 2008; Self-Report Measure for the Assessment of Emotion Regulation Skills [27 items, 9 subscales, 5-point Likert scale ("not at all" to "always")].
Change on Self-Compassion Scale (SCS-D) over multiple time points | Change from Baseline, then after six weeks and after twelve weeks
  Neff, 2003; Internationally used self-report of of self-compassion [26 items, 6 subscales, 5-point scale ("almost never" to "almost always")]. Participants will be asked to rate the items according to how often they behave in the stated manner towards themselves in difficult times.
Change on Working Alliance Inventory (WAI) between two time points | Change from six weeks after treatment to twelve weeks after
  Wilmers et al., 2008; Internationally used self-report of therapeutic alliance measuring bond, goals and tasks in psychotherapy based on feedback of patients concerning the current therapy session [online version: 12 items, 5-point Likert scale ("rarely or never" to "always")].
Change on Questionnaire Assessing the Acceptance of Unpleasant and Pleasant Emotions (Fragebogen zur Akzeptanz von Gefühlen; FrAGe) over multiple time points | Change from Baseline, then after six weeks and after twelve weeks
  Beblo et al., 2011; Self-report of the acceptance and supression of unpleasant and unpleasant emotions [32 items, 2 subscales: Pleasant and Unpleasant emotions, 6-point scale ("strongly disagree" to "strongly agree")].
Change on Positive and Negative Affect Schedule (PANAS) over multiple time points | At the beginning of every subpart of the intervention, every week up to 5 weeks
  Watson, Clark, & Tellegen, 1988; Internationally used self-report of positive and negative affect [10 items, 5-point scale ("very slightly or not at all" to "extremely")]. Participants will be asked to rate the items according to how they feel "in the current moment". The PANAS includes two subscales of global positive affect (ten items, range: 1-5) and global negative affect (10 items, range: 1-5). Only the subscale of global positive affect will be used. Subscale scores are computed with averaged item scores.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Willutzki, Prof. Dr., Study Chair — Witten/Herdecke University
Locations (1):
- Witten/Herdecke University, Witten, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Trimpop LF, Bielinski LL, Berger T, Willutzki U. Evaluation of Two Web-Based Interventions (Res-Up! and REMOTION) in Routine Outpatient Psychotherapy (Therapy Online Plus-TOP): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Mar 15;12:e41413. doi: 10.2196/41413. PMID 36920449